CLINICAL TRIAL: NCT06605495
Title: Demonstration Clinical Study of Dry Eye Disease Advantage
Brief Title: Using Dry Eye As a Disease Model, Investigators Demonstrated the Optimal Selection of Individualized Clinical Interventions and the Superiority of Dynamic Treatment Discrimination in Chinese Medicine.
Acronym: DED OSDI FBUT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuejing Lu (Other)
Responsible Party: Sponsor-Investigator, Xuejing Lu, Chief Physician of Traditional Chinese Medicine Ophthalmology, Ineye Hospital of Chengdu University of TCM, Ineye Hospital of Chengdu University of Traditional Chinese Medicine
Organization: Ineye Hospital of Chengdu University of Traditional Chinese Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024YH008
Record Dates: First submitted 2024-09-18; First posted 2024-09-20 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Dry Eye Disease (DED)
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Fumigation; Phytotherapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Chinese Medicine External Treatment Group (Active Comparator)
  Interventions: Combination Product: fumigation with Chinese medicine
- Chinese Medicine Internal Treatment Group (Oral Herbal Medicine) (Experimental)
  Interventions: Drug: Oral herbal medicine
- Western medicine treatment group (Active Comparator)
  Interventions: Drug: Modern Western Medicine

INTERVENTIONS:
Combination Product: fumigation with Chinese medicine — Eye fumigation with the Eyesight Eye Therapy,10 minutes once daily for 6 weeks.
  Arms: Chinese Medicine External Treatment Group
Drug: Oral herbal medicine — Patients were identified into the appropriate group according to the individual evidence profile, and the herbal formula under the corresponding evidence profile was taken orally as one dose of 150 ml of water twice a day for 6 weeks.
  Arms: Chinese Medicine Internal Treatment Group (Oral Herbal Medicine)
Drug: Modern Western Medicine — Referring to the Chinese Expert Consensus on Dry Eye: Treatment (2020), this course of treatment totaled 6 weeks.
  Arms: Western medicine treatment group

SUMMARY:
In this study, dry eye disease (leukoaraiosis) is used as a model disease, and the methodological system for evaluating the clinical efficacy of Chinese medicine for dry eye disease is constructed with the core of "subgrouping dynamic and static parallel group design", so as to carry out a real-world demonstration study of dry eye disease as a dominant disease in Chinese medicine treatment. The purpose of this study is to demonstrate the selection of individualized clinical interventions and the superiority of dynamic diagnosis and treatment using dry eye as a disease model. The study provides a clinical example of a subgroup-based dynamic and static parallel group design for TCM clinical research on "disease-based integrated treatment". Based on the conclusions of the efficacy evaluation study, investigators will provide real-world clinical data of dry eye syndrome for the artificial intelligence prediction of the integrated platform of individualized clinical evaluation and evidence support of Chinese medicine with multi-source data integration.

ELIGIBILITY:
Inclusion Criteria:

* Be 18-75 years of age and of any gender
* Meets Western diagnostic criteria for dry eye
* Formed consent and signed the Informed Consent Form

Exclusion Criteria:

* Those who are unable to perform a dry eye examination due to various factors
* Patients with severe diseases of the liver or renal system, or infectious eye diseases
* Those who are allergic to the medications used in this study
* Women who are pregnant or breastfeeding Mental illness or intellectual disability; Participants in clinical trials of other drugs within the last 3 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4000 (Estimated)
Dates: Start 2024-09-25 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Chinese Medical Evidence Scale | From enrollment to end of 6-week treatment
  The TCM evidence scale converts symptoms and signs into TCM evidence, and assigns 1, 2, and 3 points according to three levels of severity, with reference to the "Guiding Principles for Clinical Research on New Drugs of Traditional Chinese Medicine" and the "International TCM Clinical Practice Guidelines for Stemmed Eyes (2021-12-14)". If the points of TCM evidence are higher or unchanged after the intervention, it means that the intervention measures are ineffective or inefficient, and that patients' clinical symptoms do not improve significantly or their conditions worsen after the treatment. If the TCM syndrome score increases or remains unchanged after the intervention compared with that before treatment, it means that the intervention is ineffective or inefficient, and the patient's clinical symptoms do not improve or worsen after treatment.
Ocular Surface Disease Index | From enrollment to end of 6-week treatment
  By evaluating the points before and after the intervention treatment, if the points are lower than before the treatment, it suggests that the intervention treatment is effective, on the contrary, it indicates that the intervention is ineffective or ineffective, and the clinical symptoms of the patients do not improve significantly or worsen after the treatment.
Fluorescein Breakup Time | From enrollment to end of 6-week treatment
  Efficacy was evaluated by the values tested before and after the intervention

SECONDARY OUTCOMES:
Schirmer Ⅰ test | From enrollment to end of 6-week treatment
  Efficacy was evaluated by the values tested before and after the intervention
Height of the River of Tears | From enrollment to end of 6-week treatment
  Efficacy was evaluated by the values tested before and after the intervention
fluorescent staining of the cornea | From enrollment to end of 6-week treatment
  See the Chinese Expert Consensus on Dry Eye: Expert Consensus on Definition and Classification (2020): the cornea was divided into 4 quadrants on average, and each quadrant was scored from 0 to 3 according to the staining of sodium fluorescein, with a score of 0: no staining; 1: 1-30 punctate staining; 2: >30 punctate staining but staining not fused; and 3: fusion of the corneal punctate staining with the appearance of filaments and ulcers, etc. The final tally scores for each quadrant were summed. The efficacy was evaluated by tallying the scores detected before and after the intervention.
Classification of blepharoplasty deficiency | From enrollment to end of 6-week treatment
  The efficacy was evaluated by scoring the blepharoplasty area values detected before and after the intervention. According to the Chinese Expert Consensus on Meibomian Gland Dysfunction (2023), investigators graded the results as follows: score 0: no meibomian gland deficiency; score 1: meibomian gland deficiency ratio <1/3; score 2: meibomian gland deficiency ratio 1/3-2/3; and score 3: meibomian gland deficiency ratio >2/3.

IPD SHARING:
Plan to Share IPD: No